CLINICAL TRIAL: NCT04842695
Title: Analysis of the Effectiveness of Electroacupuncture Treatment for Urinary Incontinence in Women: A Controlled and Randomized Clinical Trial
Brief Title: Electroacupuncture Treatment for Urinary Incontinence (UI) in Women
Acronym: ELECAPUN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Electroacupuncture and UI
Record Dates: First submitted 2021-02-25; First posted 2021-04-13 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-02

CONDITIONS: Electroacupuncture; Urinary Incontinence; Women; Pelvic Floor Muscle Weakness
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Intervention Model Description: clinical study in which participants are assigned to 2 groups.Group K receive kegel´s exercise and the group A receive kegel´s exercise plus electroacupuncture in a point called R7.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- kegel´s exercise (pelvic floor exercise) (Active Comparator): A midwife/nurse works with the women according to the following protocol: 1.-identify anal sphincter, and try to raise it from chair (without adding abdominal, thigh, and buttock muscles) with a position of sitting; 2.- identify elevator ani muscle and try to raise vagina from chair (without adding abdominal, thigh, and buttock muscles) with a position of sitting, bent forward, elbows on knees; 3.- contract elevator ani muscle with a position of sitting, lying, and standing; 4.- contract anal sphincter with a position of sitting, lying, and standing. The sessions are conducted by the same midwife/nurse to women in both groups/arms to be performed by the women at home. .
  Interventions: Device: electroacupuncture group
- Electroacupuncture group (Experimental): Acupuncture point called bilateral R7 receive acupuncture with 0.25*40 mm needle with a perpendicular puncture 1.5 cun. The electrical stimulator is applied to bilateral R7, with dilatation wave 50 Hz and direct electric current of 1 milliamperes.. Each session lasts 30 minutes per day. Participants are treated 1 time per week for 12 weeks, total 12 sessions for each patient.
  Equipment:
  * Electroacupuncture device.
  * device made in China
  Interventions: Device: electroacupuncture group

INTERVENTIONS:
Device: electroacupuncture group — compare the effectiveness of electroacupuncture on point B7 plus pelvic floor exercises versus pelvic floor exercises alone in women with urinary incontinence (UI) .
  Other Names: pelvic floor exercise

SUMMARY:
The investigators have developed an investigation comparing electroacupuncture with pelvic floor exercises in female urinary incontinence (UI). It is a randomized clinical trial with 71 women with UI and two arms: 37 women received electroacupuncture with pelvic floor exercises and another arm with 34 women who only received pelvic floor exercises. The investigators evaluated the effectiveness using the International consultation on incontinence questionaire-urinary incontinence short form (ICQ-UI SF) Spanish version. The investigators also evaluated the safety of electroacupuncture in our sample.

DETAILED DESCRIPTION:
The International Continence Society defines urinary incontinence (UI) as the objectively demonstrable involuntary loss of urine. It affects women of any age. UI significantly impairs patients quality of life, limits their autonomy and reduces their self-esteem. The impairment of health-related quality of life due to UI can be even greater than that caused by some chronic diseases such as diabetes or high blood pressure.

It is common for this type of disorder to be significantly associated with depressive symptoms and feelings of anxiety, which end up affecting the physical, psychological, social, cultural and sexual levels.

UI is classified into: Stress or Effort UI (the most frequent), urge UI and mixed UI. In stress UI, involuntary urine leakage is associated with physical exertion that causes an increase in abdominal pressure; it occurs as a result of a failure in the urethral resistance mechanisms. In urge UI, the involuntary loss of urine is preceded by a compelling desire to urinate; it is due to an increase in urinary bladder contractility. In mixed UI, involuntary urine loss is associated with stress and urge incontinence.

The prevalence of UI varies according to the type of study, the definition and assessment of UI and the characteristics of the population studied (mainly age and sex, with the frequency increasing with age and in women). Worldwide, figures ranging from 5% to 72% have been published; in Spain, the available data range from 15% to 42%, the average prevalence being estimated at 40.6%. The therapeutic approach to UI can be pharmacological (anticholinergics, alpha-blockers and topical estrogens are the most commonly used agents), urological surgery, external devices (such as pessary and urethral occluder), pelvic floor exercises and stimulation by electroacupuncture.

The International Consultation on Urological Diseases recommended pelvic floor muscle training as A level evidence treating simple mild and moderate stress urinary incontinence, which curative rate varies 30% to 60%, although it is a lifelong treatment. Conservative interventions such as pelvic floor muscle training are more likely to be used than drugs or surgery while a woman is pregnant or in the postnatal period.

Pelvic floor exercises for the treatment of urinary incontinence was popularized by Arnold Kegel (1948). It has been recommended in the treatment of stress and mixed urinary incontinence, but has increasingly become part of the treatment of urge UI. It is based on two functions of the pelvic floor muscles: support of the pelvic organs, and a contribution to the urethral sphincter closure mechanism.

From the interpretation of traditional Chinese medicine, the problem of urinary incontinence may be due to a deficiency of energy or "Qi". The pelvic floor, bladder and anal sphincter need significant energy to function properly. This is why it is thought that acupuncture may be a beneficial treatment, as it may increase energy along the urinary tract. UI can be included in two syndromes depending on the signs and symptoms presented by the patient.

Our investigators work compares the effectiveness of electroacupuncture on the point R7 together with pelvic floor exercises versus pelvic floor exercises alone.

ELIGIBILITY:
Inclusion Criteria:

* Women presenting moderate-severe UI according to the ICIQ-SF questionnaire.
* Any type of urinary incontinence
* Assigned to the Torre del Mar (Malaga) health center..
* The participants gave their voluntary consent to participate in the study.

Exclusion Criteria:

* After pelvic floor operation or operation for urinary incontinence.
* Pregnancy or lactation.

  * Diagnosed neurological disease that may affect the pelvic floor.
* Grade II major genital prolapse.
* Inability to understand the messages and commands required to carry out the study procedure or answer the questionnaire.
* Women whose stay in the city is shorter than the duration of the research study.

Ages: 36 Years to 69 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 71 (Actual)
Dates: Start 2020-01-07 (Actual); Primary Completion 2021-02-05 (Actual); Study Completion 2021-02-10 (Actual)

PRIMARY OUTCOMES:
Change at 3 months in the International Consultation on Incontinence Questionnaire (ICIQ-SF) spanish version. | Change in ICIQ-SF score for each participant at 3 months
  The investigators used the ICIQ-SF questionnaire at 3 months. The investigators aimed to find a variation in the mean of the questionnaire of two or more points over the initial ICIQ-SF 0 questionnaire. The ICIQ (International Consultation on Incontinence Questionnaire) is a self-administered questionnaire that identifies individuals with urinary incontinence and the impact on quality of life.
  Any score greater than zero is considered a diagnosis of UI. Scores are from zero to 24 points. Zero points would indicate no urinary incontinence and 24 points is the highest possible score and corresponds to the highest severity of urinary incontinence.
Change at 6 months in the International Consultation on Incontinence Questionnaire (ICIQ-SF) spanish version. International Consultation on Incontinence Questionnaire (ICIQ-SF) spanish version. | change in ICIQ-SF score for each participant at 6 months.
  The investigators used the ICIQ-SF questionnaire at 6 months. The investigators aimed to find a variation in the mean of the questionnaire of two or more points over the initial ICIQ-SF 0 questionnaire. The ICIQ (International Consultation on Incontinence Questionnaire) is a self-administered questionnaire that identifies individuals with urinary incontinence and the impact on quality of life.
  Any score greater than zero is considered a diagnosis of UI. Scores are from zero to 24 points. Zero points would indicate no urinary incontinence and 24 points is the highest possible score and corresponds to the highest severity of urinary incontinence.
Change at 12 months in the International Consultation on Incontinence Questionnaire (ICIQ-SF) spanish version. | Change in ICIQ-SF score for each participant at 12 months.
  The investigators used the ICIQ-SF questionnaire at 12 months. The investigators aimed to find a variation in the mean of the questionnaire of two or more points over the initial ICIQ-SF 0 questionnaire. The ICIQ (International Consultation on Incontinence Questionnaire) is a self-administered questionnaire that identifies individuals with urinary incontinence and the impact on quality of life.
  Any score greater than zero is considered a diagnosis of UI. Scores are from zero to 24 points. Zero points would indicate no urinary incontinence and 24 points is the highest possible score and corresponds to the highest severity of urinary incontinence.

SECONDARY OUTCOMES:
appearance of adverse effects with electroacupuncture | Side effects reported for each participant through study completion, an average of 1 year. Number of Participants with pain at puncture site or hematoma or infection at puncture site during 12 months.
  The appearance of adverse effects with electroacupuncture such as pain, infection, paresthesia, hematoma or any other contingency derived from the technique applied will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Moga Lozano, doctor, Principal Investigator — Andaluz Health Service
Locations (1):
- Jose Antonio Lomeña, Málaga, Spain